CLINICAL TRIAL: NCT06359626
Title: An Open-label, Randomized, Single-dose, Oral Administration, 2-sequence, 2-period, Crossover Study to Evaluate Bioequivalence Between YHP2205 and YHR2401 in Healthy Subjects
Brief Title: Bioequivalence Study Between YHP2205 and YHR2401 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP2205-101
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Intervention Model Description: two-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence Group A (Experimental): 30 subjects, Cross-over, Single dose of YHR2401 on day 1, Single dose of YHP2205 on day 8
  Interventions: Drug: YHP2205; Drug: YHR2401
- Sequence Group B (Experimental): 30 subjects, Cross-over, Single dose of YHP2205 on day 1, Single dose of YHR2401 on day 8
  Interventions: Drug: YHP2205; Drug: YHR2401

INTERVENTIONS:
Drug: YHP2205 — Test drug: YHP2205
Drug: YHR2401 — comparator: YHR2401

SUMMARY:
A randomized, open-label, single-dose, 2-sequence, 2-period, crossover clinical trial to investigate the bioequivalence between YHP2205 and YHR2401 in healthy volunteers

DETAILED DESCRIPTION:
60 healthy subjects will be randomized to one of the 2 groups in the same ratio.

Subjects in group 1 will be administered "YHP2205" and "comparator" by cross-over design on day 1, 8

Subjects in group 2 will be administered "comparator" and "YHP2205" by cross-over design on day 1, 8.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 19 years old or older at the screening visit
* Those whose weight is > 60kg and their body mass index (BMI) shall be between 18.0 kg/m2 and 30.0 kg/m2
* Those without clinically significant congenital or chronic diseases at the screening visit and without any pathological symptom or opinion after an internal medicine examination
* Those who express their voluntary consent to participate in the trial by signing a written consent

Exclusion Criteria:

* Those who have participated in a bioequivalence study or other clinical trials and have been administered with investigational products in 6 months prior to the first administration.
* Others who are judged ineligible to participate in the trial by the principal investigator.
* Female volunteers who are pregnant, suspected to be pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-36 hours
  Area under the plasma drug concentration-time curve [AUCt] of Edoxaban
Maximum plasma concentration [Cmax] | 0-36 hours
  Maximum plasma concentration [Cmax] of Edoxaban

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] | 0-36 hours
  Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] of Edoxaban
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] | 0-36 hours
  Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] of Edoxaban
Time of peak concentration [Tmax] | 0-36 hours
  Time of peak concentration [Tmax] of Edoxaban
Terminal phase of half-life [t1/2] | 0-36 hours
  Terminal phase of half-life [t1/2] of Edoxaban

CONTACTS AND LOCATIONS:
Overall Officials: Taegon Hong, Principal Investigator — Bumin Hospital
Locations (1):
- Bumin Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No